CLINICAL TRIAL: NCT00939913
Title: N-Acetylcysteine to Prevent Contrast-Induced Nephropathy in Acute Coronary Syndromes
Brief Title: Effect of Intravenous Acetadote on Incidence of Contrast Induced Nephropathy
Acronym: NAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ochsner Health System (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Arthur G. Grant MD, Ochsner medical center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB#2006.212.A
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Nephropathy
Keywords: contrast nephropathy; intravenous n-acetlycysteine
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous N-acetlycysteine (Placebo Comparator): intravenous regimen of NAC (1,200 mg bolus followed by 200 mg/hour for 24 hours)as compared to placebo
  Acetadote provided by Cumberland Pharmaceuticals Inc.
  Interventions: Drug: intravenous NAC
- Placebo (Placebo Comparator): Study participants will be randomized to receive an intravenous regimen of NAC (1,200 mg bolus followed by 200 mg/hour for 24 hours) or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: intravenous NAC — intravenous regimen of NAC (1,200 mg bolus followed by 200 mg/hour for 24 hours)
  Arms: intravenous N-acetlycysteine
Drug: Placebo — Study participants will be randomized to receive an intravenous regimen of NAC (1,200 mg bolus followed by 200 mg/hour for 24 hours) or placebo.
  Arms: Placebo

SUMMARY:
In patients undergoing coronary angiography, the incidence of contrast induced nephropathy(CIN)varies widely and ranges from < 5% in the lowest risk patients, to nearly 50% in the highest risk patients. Prior data has shown oral n-acetyl cysteine (NAC) to be effective in reducing the incidence of CIN.Due to extensive first pass metabolism, the bioavailability of oral NAC is poor and ranges from 4%-10%. We hypothesize that the incidence of CIN will be reduced in patients with ACS who undergo PCI by the prophylactic administration of intravenous NAC.

This is a prospective, randomized, double-blind, placebo-controlled single center clinical trial designed to evaluate the effects of intravenous NAC on patients with acute coronary syndromes (ACS)undergoing coronary angiography and/or percutaneous coronary intervention (PCI). The medication Acetadote is provided by Cumberland Pharmaceuticals Inc (www.cumberlandpharma.com).

Patients will be excluded if they have end-stage renal disease requiring dialysis,known hypersensitivity to NAC or a history of life-threatening contrast reaction. Primary end-point is incidence of CIN. Secondary end-points are in-hospital mortality,30-day mortality,duration of hospitalization and change in serum cystatin C level.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Hospitalized with a primary diagnosis of acute coronary syndrome.
3. Scheduled for coronary angiography or intervention during the current hospitalization.

Exclusion Criteria:

1. Have end-stage renal disease (ESRD) requiring dialysis.
2. Have a known hypersensitivity to NAC.
3. Have a history of life-threatening contrast reaction. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of CIN | 48-72 hours

SECONDARY OUTCOMES:
in-hospital mortality | 30 days
30 day mortality | 30 days
duration of hospitalization | 30 days
serum cystatin C | 48-72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Jaffery Z, Verma A, White CJ, Grant AG, Collins TJ, Grise MA, Jenkins JS, McMullan PW, Patel RA, Reilly JP, Thornton SN, Ramee SR. A randomized trial of intravenous n-acetylcysteine to prevent contrast induced nephropathy in acute coronary syndromes. Catheter Cardiovasc Interv. 2012 May 1;79(6):921-6. doi: 10.1002/ccd.23157. Epub 2011 Nov 30. PMID 21542122